CLINICAL TRIAL: NCT01703481
Title: A Phase 1 Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-42756493, a Pan-Fibroblast Growth Factor Receptor (FGFR) Tyrosine Kinase Inhibitor, in Subjects With Advanced or Refractory Solid Tumors or Lymphoma
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-42756493 in Adult Participants With Advanced or Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100845; 42756493EDI1001 (Other: Janssen Research & Development, LLC); 2012-000697-34 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-10-10 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Tumor or Lymphoma
Keywords: Tumor; Fibroblast Growth Factor Receptor (FGFR); Non-Small Cell Lung Cancer (NSCLC); Small Cell Lung Cancer (SCLC); JNJ-42756493
MeSH Terms: conditions — Neoplasms; Lymphoma; Acrocephalosyndactylia; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1 (Experimental): Dose Escalation, Part 1: Participants will be enrolled in sequential cohorts to determine recommended Phase 2 doses (RP2D).
  Interventions: Drug: JNJ-42756493: Part 1
- Part 2 (Experimental): Dose Confirmation, Part 2: Tumor biopsy cohorts will confirm RP2D.
  Interventions: Drug: JNJ-42756493: Part 2
- Part 3, Cohort A (Experimental): First dose expansion, Part 3: Participants with squamous non-small cell lung cancer.
  Interventions: Drug: JNJ-42756493: Part 3
- Part 3, Cohort B (Experimental): First dose expansion, Part 3: Participants with small cell lung cancer.
  Interventions: Drug: JNJ-42756493: Part 3
- Part 3, Cohort C (Experimental): First dose expansion, Part 3: Participants with breast cancer.
  Interventions: Drug: JNJ-42756493: Part 3
- Part 3, Cohort D (Experimental): First dose expansion, Part 3: Participants with solid tumors (consisting of one of the following: gastric, head and neck, lung adenocarcinoma, urothelial, glioblastoma multiforme [GBM], ovarian or prostate).
  Interventions: Drug: JNJ-42756493: Part 3
- Part 4, Cohort E (Experimental): Second dose expansion, Part 4: Participants with non-small cell lung cancer.
  Interventions: Drug: JNJ-42756493: Part 4
- Part 4, Cohort F (Experimental): Second dose expansion, Part 4: Participants with solid tumors (consisting of one of the following: breast, urothelial, GBM).
  Interventions: Drug: JNJ-42756493: Part 4

INTERVENTIONS:
Drug: JNJ-42756493: Part 1 — Participants will receive 0.5 mg (starting dose) capsule of JNJ-42756493 orally (by mouth) once daily on Day 1 of Cycle 1. Dose of the study medication will be escalated sequentially till the dose limiting toxicity is achieved to determine the recommended part 2 doses (RP2D).
  Arms: Part 1
Drug: JNJ-42756493: Part 2 — Participants will receive JNJ-42756493 at the RP2D or below RP2D (maximum tolerated dose from Part 1) orally once daily on a 21 days cycle to confirm RP2D (in Part 2).
  Arms: Part 2
Drug: JNJ-42756493: Part 3 — Participants will receive JNJ-42756493 at first RP2D of 9 mg daily in Part 3 orally once daily on a 21 days cycle.
  Arms: Part 3, Cohort A; Part 3, Cohort B; Part 3, Cohort C; Part 3, Cohort D
Drug: JNJ-42756493: Part 4 — Participants will receive JNJ-42756493 second RP2D of 10 mg intermittent dosing in Part 4 (with option to increase to 12 mg intermittent dosing based on phosphate level), orally on an intermittent schedule of daily for 7 days followed by 7 days off with a 28-day cycle.
  Arms: Part 4, Cohort E; Part 4, Cohort F

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (study of what the body does to a drug), and pharmacodynamics (study of what a drug does to the body) of JNJ-42756493, a pan-fibroblast growth factor receptor (FGFR) tyrosine kinase inhibitor, in adult participants with advanced or refractory solid tumors or lymphoma.

DETAILED DESCRIPTION:
This is a first-in-human, non-randomized (individuals will not be assigned by chance to study treatments), open-label (individuals will know the identity of study treatments), multicenter (more than 1 hospital work on a study), Phase 1 study. The study consists of 4 parts. Part 1 is the dose-escalation phase, which will be guided by pharmacokinetics, pharmacodynamics and safety. In part 1, safe and biologically active Phase 2 doses (recommended Phase 2 doses [RP2D]) for JNJ-42756493 will be primarily assessed. Participants will be enrolled in sequential cohorts (first cohort will receive the starting dose and subsequent cohorts will receive increased doses of JNJ-42756493). Part 2 is the Dose Confirmation Phase, which consists of a pre and post treatment tumor biopsy cohorts to confirm the RP2D based on the pharmacodynamic effect of JNJ-42756493 on fibroblast growth factor receptor (FGFR) signaling pathway in tumor. Part 3 is the first Dose Expansion Phase, which is designed to evaluate inclusion biomarkers and preliminary clinical activity at the first RP2D. It consists of 4 expansion cohorts, 1 each for squamous cell lung cancer, small cell lung cancer, breast cancer, other solid tumors (Cohorts A, B, C, and D). Part 4 is the second Dose Expansion Phase, which is designed to evaluate inclusion biomarkers and preliminary clinical activity at the second RP2D. Biomarker eligibility has also been refined based on emerging data. It consists of 2 expansion cohorts, Cohort E for non-small cell lung cancer and Cohort F for select solid tumors including breast, urothelial, GBM, ovarian, head & neck, esophageal, gastric, and cholangiocarcinoma (Cohorts E and F). Enrollment of some cohorts may be discontinued due to lack of enrollment or for futility. The study is estimated to take approximately 48 months to complete. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed: solid malignancy or lymphoma that is metastatic or unresectable, and for which standard curative treatment is no longer effective (Part 1); any type of advanced or refractory solid malignancy (excluding lymphoma) that is metastatic or unresectable and for which standard curative treatment is no longer effective (Part 2); advanced or refractory squamous non-small cell lung cancer (Cohort A, Part 3), advanced or refractory small cell lung cancer (Cohort B, Part 3), advanced or refractory breast cancer (Cohort C, Part 3), any type of advanced or refractory solid malignancy (excluding lymphoma) ([consisting of one of the following: gastric, head and neck, lung adenocarcinoma, urothelial, glioblastoma multiforme (GBM), ovarian or prostate]) (Cohort D, Part 3), advanced or refractory non small cell lung cancer(Cohort E, Part 4), any type of advanced or refractory solid malignancy (consisting of one of the following: Breast, Urothelial, GBM, Ovarian, Head & Neck, Esophageal, Gastric, and Cholangiocarcinoma) (Cohort F, Part 4)
* Eastern Cooperative Oncology Group performance status score 0 or 1
* Adequate bone marrow, liver, and renal function within the 14 days prior to Day 1 of Cycle 1 of study drug up until pre-dose of Cycle 1
* Magnesium within 0.85 to 1.25 * institutional normal limits, Sodium greater than or equal to 130 milli equivalent per liter, Potassium within institutional normal limits (within 14 days prior to Day 1 of Cycle 1 up until pre-dose of Cycle 1)

Exclusion Criteria:

* Chemotherapy, targeted therapies, radiotherapy, immunotherapy, or treatment with an investigational anticancer agent within 2 weeks or at least 5 half-lives of the drug, whichever is longer and up to a maximum of 4 weeks (in the case of nitrosoureas and mitomycin C within 6 weeks) before the first administration of study drug. Localized radiation therapy and ongoing luteinizing hormone-releasing hormone (LHRH) agonists, bisphosphonates and denosumab, are permitted
* Participants with GBM can be enrolled 2 weeks after last treatment
* History or current condition of uncontrolled cardiovascular disease
* Participants with persistent phosphate greater than upper limit of normal during screening (within 14 days prior to Day 1 of Cycle 1 up until pre-dose of Cycle 1) and despite medical management of phosphate levels
* Participants taking medications known to have a significant risk of causing QTc prolongation and Torsades de Pointes
* Left ventricular ejection fraction (LVEF) less than 50 percent as assessed by echocardiography (or multi-gated acquisition) performed at screening
* Any medical condition that requires intact wound healing capacity and is expected to endanger participant safety if wound healing capacity would be severely reduced during administration of the investigational agent
* Participants not recovered from reversible toxicity of prior anticancer therapy (except toxicities which are not clinically significant such as alopecia, skin discoloration, or Grade 1 neuropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Tolerated Dose (MTD) of JNJ-42756493 | Up to Part 1 Day 84 (Cycle 4, Day 21)
  The maximum tolerated dose as determined in Part 1 of the study will be used as the recommended dose for Part 2, 3 and Part 4.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-42756493 | Up to Part 4 Day 84 (Cycle 4, Day 21)
  The Cmax is the maximum observed plasma concentration.
Minimum Observed Plasma Concentration (Cmin) of JNJ-42756493 | Up to Part 4 Day 84 (Cycle 4, Day 21)
  The Cmin is the minimum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-42756493 | Up to Part 4 Day 84 (Cycle 4, Day 21)
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Up to Part 4 Day 84 (Cycle 4, Day 21)
  The AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval (24 hour). It is used to characterize drug absorption.
Elimination Half Life of JNJ-42756493 | Up to Part 4 Day 84 (Cycle 4, Day 21)
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Apparent Volume of Distribution at Steady-State (Vss) of JNJ-42756493 | Up to Part 4 Day 84 (Cycle 4, Day 21)
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steady-state, which is estimated by (D/AUC[0-infinity])*(AUMC[0-infinity])/AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time.
Total Clearance of JNJ-42756493 | Up to Part 4 Day 84 (Cycle 4, Day 21)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Total clearance of drug is calculated as dose divided by AUCtau at steady-state.
Accumulation Index (AI) of JNJ-42756493 | Up to Part 4Day 84 (Cycle 4, Day 21)
  Accumulation index is calculated by Cmax on Day 1 of Cycle 2/Cmax on Day 1 of Cycle 1 and/or AUCtau on Day 1 of Cycle 2/AUCtau on Day 1 of Cycle 1, where tau is the length of the dosing interval (24 hour).
Number of Participants With Objective Tumor Response | Up to Part 4 Day 84 (Cycle 4, Day 21)
  Objective response based on assessment of confirmed Complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST). CR defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than 10 millimeter (mm). PR defined as at least 30 percent (%) decrease in sum of the diameters of the target lesions taking as reference the Baseline sum diameters. Confirmed responses are those that persist on repeat imaging study for at least 4 weeks after initial documentation of response.
Progression Free Survival (PFS) | Up to Part 4 Day 84 (Cycle 4, Day 21)
  Progression free survival is the time period from start of study medication till the disease progression or death, whichever occurs first.
Duration of Objective Response | Up to Part 4 Day 84
  Duration of objective response is time interval from the first date that criteria for complete response or partial response are met to the first date of progression of disease.
Number of Participants With an Adverse Event | Up to Part 4 Day 84 (Cycle 4, Day 21)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (37):
- United States (23):
  - Birmingham, Alabama
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Sacramento, California
  - Santa Monica, California
  - Denver, Colorado
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Goshen, Indiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Tyler, Texas
  - Fairfax, Virginia
- France (7):
  - Bordeaux
  - Caen
  - Dijon
  - Lyon
  - Marseille
  - Saint-Herblain
  - Villejuif
- Spain (7):
  - Badalona
  - Barcelona
  - Madrid
  - Málaga
  - Pamplona
  - Seville
  - Valencia

REFERENCES:
- [Result] Tabernero J, Bahleda R, Dienstmann R, Infante JR, Mita A, Italiano A, Calvo E, Moreno V, Adamo B, Gazzah A, Zhong B, Platero SJ, Smit JW, Stuyckens K, Chatterjee-Kishore M, Rodon J, Peddareddigari V, Luo FR, Soria JC. Phase I Dose-Escalation Study of JNJ-42756493, an Oral Pan-Fibroblast Growth Factor Receptor Inhibitor, in Patients With Advanced Solid Tumors. J Clin Oncol. 2015 Oct 20;33(30):3401-8. doi: 10.1200/JCO.2014.60.7341. Epub 2015 Aug 31. PMID 26324363
- [Derived] Valade E, Dosne AG, Xie H, Kleiman R, Li LY, Perez-Ruixo JJ, Ouellet D. Assessment of the effect of erdafitinib on cardiac safety: analysis of ECGs and exposure-QTc in patients with advanced or refractory solid tumors. Cancer Chemother Pharmacol. 2019 Sep;84(3):621-633. doi: 10.1007/s00280-019-03896-1. Epub 2019 Jul 6. PMID 31280362
- [Derived] Bahleda R, Italiano A, Hierro C, Mita A, Cervantes A, Chan N, Awad M, Calvo E, Moreno V, Govindan R, Spira A, Gonzalez M, Zhong B, Santiago-Walker A, Poggesi I, Parekh T, Xie H, Infante J, Tabernero J. Multicenter Phase I Study of Erdafitinib (JNJ-42756493), Oral Pan-Fibroblast Growth Factor Receptor Inhibitor, in Patients with Advanced or Refractory Solid Tumors. Clin Cancer Res. 2019 Aug 15;25(16):4888-4897. doi: 10.1158/1078-0432.CCR-18-3334. Epub 2019 May 14. PMID 31088831